CLINICAL TRIAL: NCT03849274
Title: Effectiveness of a Combined Adequate Pressure and Silicone Intervention in Comparison With Conventional Pressure for Hypertrophic Scar Treatment
Brief Title: SMART Dressing for Hypertrophic Scar Treatment Post-Total Knee/Hip Arthroplasty
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr. Ho Ki Wai, Clinical Professional Consultant, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CUHK_2018.487-T
Record Dates: First submitted 2019-02-11; First posted 2019-02-21 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Knee Arthropathy; Hip Arthropathy; Hypertrophic Scar
Keywords: Knee Arthropathy; Hip Arthopathy; Hypertrophic Scar; Smart Scar Care Pad; Pressure Garment
MeSH Terms: conditions — Cicatrix, Hypertrophic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All subjects will be asked to removed all the treatment materials before they entered the assessment rooms to ensure the blinding of the assessor. The ultrasound data will be processed and analysed by blinded analysts.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Smart Scar Care Pad+Pressure Garment (Experimental): For experiment group, subject will be intervened by SSCP plus PG
  Interventions: Combination Product: Smart Scar Care Pad=Pressure Garment; Device: Pressure Garment
- Pressure Garment (Active Comparator): For control group, subject will be intervened by conventional PG only
  Interventions: Device: Pressure Garment
- Non-eligible patients (with VSS less than 4) (No Intervention): Non-eligible subjects with VSS less than 4 will be followed up for 6 months and assessment results will be recorded.

INTERVENTIONS:
Combination Product: Smart Scar Care Pad=Pressure Garment — Smart Scar Care Pad (SSCP) + conventional Pressure Garment in the management of HS in adult with total hip replacement (THR) and total knee replacement (TKR)
  Arms: Smart Scar Care Pad+Pressure Garment
Device: Pressure Garment — Conventional Pressure Garment (PG) alone in the management of HS in adult with total hip replacement (THR) and total knee replacement (TKR)
  Arms: Pressure Garment; Smart Scar Care Pad+Pressure Garment

SUMMARY:
Pressure therapy (PT) and silicone therapy are recommended as first-line non-invasive treatment for Hypertrophic Scar (HS), yet the effectiveness of the combination of these two treatments through an RCT trial has not been established yet. This study aims to examine the effectiveness of the combination of adequate pressure therapy and silicone gel sheeting implemented by Smart Scar Care Pad (SSCP) + conventional Pressure Garment (PG) versus conventional Pressure Garment (PG) alone in the management of HS in adult with total hip replacement (THR) and total knee replacement (TKR). This study also aims to find out the prevalence of hypertrophic scar among patients with THR and TKR. This study is a randomised controlled trial with two parallel arms, with allocation ratio (Experimental: Control) of 1: 1 in order to establish the superiority of SSCP + PG over PG. Subjects with hypertrophic scar will be randomly assigned to either treatment or control group. The subjects in the treatment group will be provided with the SSCP and PG for treatment, whereas the subjects in the control group will be prescribed only the PG. The treatment will last for a total of 6 months. A variety of objective outcome measures will be used to analysis the treatment effect.

DETAILED DESCRIPTION:
Hypertrophic scar (HS) is a challenging yet common complication of dermal injuries such as burns, surgeries, and trauma. It is characterized as a raised, rigid, hyper-vascular, and abnormally pigmented scar confined within the border of the initial injury. The induced aesthetic defect and impaired physical function could adversely affect quality of life.1 Pressure therapy (PT) and silicone therapy are recommended as first-line non-invasive treatments HS.

Recent reviews suggested PT was able to decrease scar height and erythema3,4. The inconclusive outcome results from fact that seldom research address the issue of adequate pressure dosage, which is essential for the treatment effect of PT. It is recommended that an interface pressure of 15-25 mmHg should be given and maintained through a 23 hrs/day wearing regime in order to achieve optimal treatment outcomes5. However, maintaining adequate pressure dosage through pressure garment alone is usually uncomfortable and sometimes impossible, especially over bodily concave area. Therefore, pressure inserts are used in conjunction with pressure garment to increase local pressure6. Despite the documented use of pressure inserts in various journals, pressure garment alone remains the mainstream treatment for hypertrophic scar.

Cochrane review conducted on silicone gel sheet (SGS) revealed SGS's ability in reducing scar thickness and improving scar color, but insufficient data on its effect on scar pliability5. SGS are commonly used to occlude and provide hydration to scar tissues.5, 6 They are mainly used for small scars or surgical scars. They are generally costly and thin in physical form, rendering them incapable of exerting sufficient pressure.

The joint effectiveness of these two treatment modalities in scar management is always drawing the interests from researchers. Various studies reported that enhanced effectiveness could be achieved through the combination of PT and SGS especially in terms of scar pliability, though all subjectively measured6-8. Therefore, there is an urging need to establish the effectiveness of the combination of these two treatments through an RCT.

In order to address the adequate pressure as well as the silicone gel sheeting effect at the same time, a newly invented insert material, the Smart Scar Care Pad (SSCP), is adopted in this study as treatment modality. The Smart Scar Care Pad is especially designed with a rubbery silicone stiffener layer and medical grade silicone gel lining layer underneath. The medical grade silicone gel lining layer underneath serves as the occlusion layer. The rubbery silicone stiffener layer is designed with numerous studs. By cutting the individual studs into gradient height, the Smart Scar Care Pad (SSCP), creates tailor made localized pressure under pressure garment. Studs are also aligned in honey cone style in order to maximize conformability over different bodily contours. In that case, the Smart Scar Care Pad (SSCP) not only increases local pressure but also provides occlusion to HS tissue.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (age over 18 years old) undergoing TKR and THR within 6 weeks;
2. Adult who is able to provide written consent, is cooperative and compliant with the treatment and assessment regime;
3. The Vancouver Scar Scale (VSS) will be used to screen candidates for the study.10 Isolated scars with a total score of 4 or higher and the score of each item equal to or greater than 1 will be included.

   Exclusion Criteria:
4. The HS area has an open wound or infection, or HS area is local flap or skin graft area;
5. The HS area intends to be treated with steroid injections or other interventions (such as traditional Chinese medicine or laser therapy)
6. The patients with co-morbidities that might affect their compliance to treatment such as dermatological disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Changes from baseline hypertrophic Scar Thickness at 1 months post-surgical to total knee/hip arthroplasty | 1 month post total knee/hip arthroplasty operation
  Using an ultrasound machine, thickness of scar is aggregately measured to the average of 3 points: the center of the inner ring, 5 mm on both side of the centre point, which reflected the points of circumference of the selected scar sites.
Changes from baseline hypertrophic Scar Thickness at 3 months post-surgical to total knee/hip arthroplasty | 3 month post total knee/hip arthroplasty operation
  Using an ultrasound machine, thickness of scar is aggregately measured to the average of 3 points: the center of the inner ring, 5 mm on both side of the centre point, which reflected the points of circumference of the selected scar sites.
Changes from baseline hypertrophic Scar Thickness at 6 months post-surgical to total knee/hip arthroplasty | 6 month post total knee/hip arthroplasty operation
  Using an ultrasound machine, thickness of scar is aggregately measured to the average of 3 points: the center of the inner ring, 5 mm on both side of the centre point, which reflected the points of circumference of the selected scar sites.

SECONDARY OUTCOMES:
Changes of scar vascularity and pigmentation at 1 month post-surgical to total knee/hip arthroplasty | 1 month post total knee/hip arthroplasty operation
  Hypertrophic scar vascularity and pigmentation will be measured using the Dermlite Foto II Pro (3GEN Inc., San Juan Capistrano, CA, USA).
Changes of scar vascularity and pigmentation at 3 months post-surgical to total knee/hip arthroplasty | 3 months post total knee/hip arthroplasty operation
  Hypertrophic scar vascularity and pigmentation will be measured using the Dermlite Foto II Pro (3GEN Inc., San Juan Capistrano, CA, USA).
Changes of scar vascularity and pigmentation at 6 month post-surgical to total knee/hip arthroplasty | 6 month post total knee/hip arthroplasty operation
  Hypertrophic scar vascularity and pigmentation will be measured using the Dermlite Foto II Pro (3GEN Inc., San Juan Capistrano, CA, USA).
Changes of scar elasticity at 1 month post-surgical to total knee/hip arthroplasty | 1 month post total knee/hip arthroplasty operation
  Hypertrophic scar elasticity will be measured using the DermaLab Combo (Cortex Technology, Hadsund, Denmark)
Changes of scar elasticity at 3 months post-surgical to total knee/hip arthroplasty | 3 months post total knee/hip arthroplasty operation
  Hypertrophic scar elasticity will be measured using the DermaLab Combo (Cortex Technology, Hadsund, Denmark)
Changes of scar elasticity at 6 months post-surgical to total knee/hip arthroplasty | 6 months post total knee/hip arthroplasty operation
  Hypertrophic scar elasticity will be measured using the DermaLab Combo (Cortex Technology, Hadsund, Denmark)
Changes of range of motion (ROM) of knee joint or hip joint at 1 month post-surical to total knee/hip arthroplasty | 1 month post total knee/hip arthroplasty operation
  It describes the joint movement range. Physical therapist will manually bend and straighten patients' knee, passively moving legs .
Changes of range of motion (ROM) of knee joint or hip joint at 3 months post-surical to total knee/hip arthroplasty | 3 months post total knee/hip arthroplasty operation
  It describes the joint movement range. Physical therapist will manually bend and straighten patients' knee, passively moving legs .
Changes of range of motion (ROM) of knee joint or hip joint at 6 months post-surical to total knee/hip arthroplasty | 6 months post total knee/hip arthroplasty operation
  It describes the joint movement range. Physical therapist will manually bend and straighten patients' knee, passively moving legs .
Changes of circumference measurement of knee joint or hip joint at 1 month post-surgical to total knee/hip arthroplasty | 1 month post-surgical to total knee/hip arthroplasty
  It describes the circumference of joint in centimeter units.
Changes of circumference measurement of knee joint or hip joint at 3 months post-surgical to total knee/hip arthroplasty | 3 months post-surgical to total knee/hip arthroplasty
  It describes the circumference of joint in centimeter units.
Changes of circumference measurement of knee joint or hip joint at 6 months post-surgical to total knee/hip arthroplasty | 6 months post-surgical to total knee/hip arthroplasty
  It describes the circumference of joint in centimeter units.
Changes of pain/itchiness sensation at 1 month post-surgical to total knee/hip arthroplasty | 1 month post-surgical to total knee/hip arthroplasty
  Numerical rating scale (NRS) will be used to measure itchiness and pain. Patient are asked to point to the number on the Numeric Rating Scale that best represents the intensity of their pain NOW. The scale have a scale ranges from 0 to 10, with higher the number considering the worse possible pain/itchiness sensation.
Changes of pain/itchiness sensation at 3 months post-surgical to total knee/hip arthroplasty | 3 months post-surgical to total knee/hip arthroplasty
  Numerical rating scale (NRS) will be used to measure itchiness and pain. Patient are asked to point to the number on the Numeric Rating Scale that best represents the intensity of their pain NOW. The scale have a scale ranges from 0 to 10, with higher the number considering the worse possible pain/itchiness sensation.
Changes of pain/itchiness sensation at 6 months post-surgical to total knee/hip arthroplasty | 6 months post-surgical to total knee/hip arthroplasty
  Numerical rating scale (NRS) will be used to measure itchiness and pain. Patient are asked to point to the number on the Numeric Rating Scale that best represents the intensity of their pain NOW. The scale have a scale ranges from 0 to 10, with higher the number considering the worse possible pain/itchiness sensation.
Changes of The 36-Item Short Form Health Survey (SF-36) index at 1 month post-surgical to total knee/hip arthroplasty | 1 month post-surgical to total knee/hip arthroplasty
  The 36-Item Short Form Health Survey (SF-36) will be used to measure the health related Quality of Life. The SF-36 has eight scaled scores; the scores are weighted sums of the questions in each section. Scores range from 0 - 100. Lower scores = more disability, higher scores = less disability.
Changes of The 36-Item Short Form Health Survey (SF-36) index at 3 months post-surgical to total knee/hip arthroplasty | 3 months post-surgical to total knee/hip arthroplasty
  The 36-Item Short Form Health Survey (SF-36) will be used to measure the health related Quality of Life. The SF-36 has eight scaled scores; the scores are weighted sums of the questions in each section. Scores range from 0 - 100. Lower scores = more disability, higher scores = less disability.
Changes of The 36-Item Short Form Health Survey (SF-36) index at 6 months post-surgical to total knee/hip arthroplasty | 6 months post-surgical to total knee/hip arthroplasty
  The 36-Item Short Form Health Survey (SF-36) will be used to measure the health related Quality of Life. The SF-36 has eight scaled scores; the scores are weighted sums of the questions in each section. Scores range from 0 - 100. Lower scores = more disability, higher scores = less disability.
Changes of treatment satisfaction value at 1 month post-surgical to total knee/hip arthroplasty | 1 month post-surgical to total knee/hip arthroplasty
  Numerical rating scale (NRS) will be used to measure treatment satisfaction. Patient are asked to point to the number on the Numeric Rating Scale that best represents the intensity of their pain NOW. The scale have a scale ranges from 0 to 10, with higher the number considering the better treatment satisfaction.
Changes of treatment satisfaction value at 3 months post-surgical to total knee/hip arthroplasty | 3 months post-surgical to total knee/hip arthroplasty
  Numerical rating scale (NRS) will be used to measure treatment satisfaction. Patient are asked to point to the number on the Numeric Rating Scale that best represents the intensity of their pain NOW. The scale have a scale ranges from 0 to 10, with higher the number considering the better treatment satisfaction.
Changes of treatment satisfaction value at 6 months post-surgical to total knee/hip arthroplasty | 6 months post-surgical to total knee/hip arthroplasty
  Numerical rating scale (NRS) will be used to measure treatment satisfaction. Patient are asked to point to the number on the Numeric Rating Scale that best represents the intensity of their pain NOW. The scale have a scale ranges from 0 to 10, with higher the number considering the better treatment satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Orthopaedics & Traumatology, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided